CLINICAL TRIAL: NCT02856516
Title: Plasma Glucose and Insulin Response to Three Oral Nutrition Supplements in Persons With Type 2 Diabetes Mellitus
Brief Title: Glycemic Response to Three Oral Nutrition Supplements in Persons With Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 15.11.US.HCN
Record Dates: First submitted 2016-08-02; First posted 2016-08-05 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-07

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Boost Glucose Control (A) (Experimental): Nutritional beverage (Oral Nutrition Supplement) designed for oral consumption in people with Diabetes.
  Interventions: Other: Boost Glucose Control (A)
- Boost Glucose Control (B) (Experimental): Nutritional beverage (Oral Nutrition Supplement) designed for oral consumption in people with Diabetes.
  Interventions: Other: Boost Glucose Control (B)
- Boost Original (Active Comparator): Nutritional beverage (Oral Nutrition Supplement) designed for oral consumption.
  Interventions: Other: Boost Original

INTERVENTIONS:
Other: Boost Glucose Control (A) — Oral nutrition supplement
  Arms: Boost Glucose Control (A)
Other: Boost Glucose Control (B) — Oral nutrition supplement
  Arms: Boost Glucose Control (B)
Other: Boost Original — Oral nutrition supplement
  Arms: Boost Original

SUMMARY:
This will be a randomized, cross-over design. Subjects will be randomized to one of three interventions on three separate study days, 1 week apart.

DETAILED DESCRIPTION:
Following consent, subjects will be randomized to one of three arms. After an overnight fast an intravenous line will be placed for blood withdrawal. The subject will then consume the randomly assigned intervention. Blood samples for glucose and insulin levels will be drawn at specified intervals after the product has been consumed.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-75 yrs
* Type 2 diabetes controlled with diet or diet and oral agent, with the exception of sulfonylureas such as glimepiride (Amaryl), glipizide (Glucotrol/Glucotrol XL) and glyburide (DiaBeta, Micronase, (Glynase Prestabs); meglitinides such as reaglinide (Prandin) and nateglinide (Starlix); and alphaglucosidase inhibitors such as acarbose (Precose) and miglitol (Glyset)
* Hemoglobin A1C less than 9.0%
* Fasting blood glucose less than 180 mg

Exclusion Criteria:

* Abnormal thyroid function
* Creatinine >2.0 mg/dL
* Potassium <3.5 mEq/L
* Gastrointestinal disease: ulcer, gastritis, diarrhea, gastroparesis, vomiting
* Currently unstable diabetes or under treatment for cancer, heart disease, renal disease
* Unable to give informed consent or follow instructions
* Current insulin therapy or insulin therapy within the past month
* Patients who are pregnant
* Allergies to milk, soy or any component of the test product
* Patient who in the Investigators assessment cannot be expected to comply with treatment
* Currently participating or having participated in another clinical trial.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-07; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Area under the blood glucose curve (AUC 0-240) | Baseline, 10, 20, 30, 60, 90, 120, 150, 180, 210 and 240 minutes

SECONDARY OUTCOMES:
Area under the insulin curves (AUC 0-240) | Baseline, 10, 20, 30, 60, 90, 120, 150, 180, 210 and 240 minutes
Insulinogenic index (Ins30/(Glu30) | Baseline, 10, 20, 30, 60, 90, 120, 150, 180, 210 and 240 minutes
AUC (0-30min) for insulin | Baseline, 10, 20, 30, 60, 90, 120, 150, 180, 210 and 240 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Joel Neutel, MD, Principal Investigator — Orange County Research Center
Locations (1):
- Orange County Research Center, Tustin, California, United States

IPD SHARING:
Plan to Share IPD: No
Data will be presented in a peer reviewed manuscript